CLINICAL TRIAL: NCT05180292
Title: Acute Hemodynamic Response to Carvedilol in Predicting Survival in Acute on Chronic Liver Failure Patients - A Pilot Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-11
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute on Chronic Liver failure (Experimental)
  Interventions: Drug: Carvedilol 12.5 MG

INTERVENTIONS:
Drug: Carvedilol 12.5 MG — Carvedilol 12.5 mg

SUMMARY:
Various parameters will be assessed during the procedure before and after 1 hour of 12.5 mg carvedilol such as HVPG (WHVP - FHVP), SVR, heart rate, cardiac output, cardiac index, Blood pressure (systolic, diastolic and mean), SpO2. Routine treatment of the patients will be continued as per the Institute protocol. These patients will be assessed for the liver transplant free survival at 28 days and complications [PHT related bleed, AKI, infections, HE] within 90 days; transplant-free survival rate at 90 days; evolution of the AARC score for 2 wk.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of ACLF (APASL criteria) - jaundice (serum bilirubin ≥ 5 mg/dL and coagulopathy (INR ≥ 1.5) complicated within 4 weeks by clinical ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease/cirrhosis,
2. Age 18-70 yrs
3. Baseline HVPG ≥ 12 mmHg.

Exclusion Criteria:

1. Contraindications to NSBB (heart rate < 65 /min, BP < 110/65 mm Hg, asthma, heart failure),
2. Portal Vein Thrombosis,
3. Hepatocellular carcinoma,
4. HVOTO,
5. HE grades 2-4,
6. NSBB therapy within 5 days,
7. Pregnancy,
8. Lactation,
9. Planned for LT in the next 12 weeks
10. No consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver transplant free survival | Day 28

SECONDARY OUTCOMES:
Complications [PHT related bleed, AKI, infections, HE] within 90 days | 90 days
Liver transplant-free survival rate | 90 days
Correlation with evolution of AARC score | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No